CLINICAL TRIAL: NCT01703507
Title: Phase I Study of Ipilimumab Combined With Whole Brain Radiation Therapy or Radiosurgery for Melanoma Patients With Brain Metastases
Brief Title: Phase I Study of Ipilimumab Combined With Whole Brain Radiation Therapy or Radiosurgery for Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12P.314; 2012-43 (Other: CCRRC); JT 2988 (Other: JeffTrial Number)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma; Tumors Metastatic to Brain
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Ipilimumab and Whole Brain Radiation Therapy) (Experimental): Patients receive ipilimumab IV over 90 minutes once in weeks 1, 4, 7, and 10. Patients also undergo WBRT 5 days a week in weeks 1-2.
  Interventions: Drug: Ipilimumab; Radiation: Whole-Brain Radiation Therapy (WBRT)
- Arm B (Ipilimumab and Stereotactic Radiosurgery) (Experimental): Patients receive ipilimumab IV over 90 minutes as in Arm A. Patients also undergo SRS on day 1 in week 1.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Drug: Ipilimumab — Given IV
  Other Names: MDX-010; MDX-101; Yervoy
Radiation: Whole-Brain Radiation Therapy (WBRT) — Undergo WBRT
  Other Names: WBRT; Whole-brain radiotherapy
  Arms: Arm A (Ipilimumab and Whole Brain Radiation Therapy)
Radiation: Stereotactic Radiosurgery (SRS) — Undergo SRS
  Arms: Arm B (Ipilimumab and Stereotactic Radiosurgery)

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab when given together with whole brain radiation therapy or stereotactic radiosurgery in treating patients with melanoma with brain metastases. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some block the ability of the tumor to grow and spread. Others find Tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy, such uses high-energy x-rays and other types of radiation to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells. Giving ipilimumab together with whole-brain radiation therapy or stereotactic radiosurgery may kill more tumor cells.

DETAILED DESCRIPTION:
Melanoma patients with brain metastases have a very poor outcome. Most patients with brain metastases will die from CNS related death. Radiation therapy is an effective treatment for patients with brain metastases for symptom palliation and survival benefit. Patients with multiple metastases are typically treated with whole brain radiation treatment (WBRT). For patients with a few metastases, stereotactic radiosurgery (SRS) alone can be used as an alternative. CTLA-4 (Cytotoxic T-Lymphocyte Antigen 4) antibody, Ipilimumab has shown efficacy in metastatic melanoma and unresectable melanoma. Treatment with high doses of radiation therapy would result in tumor cell death, releasing tumor debris and liberating potential tumor antigens. We hypothesize that combining radiation therapy with Ipilimumab will facilitate immune recognition of these novel tumor-specific antigens, yielding a synergistic effect. Further, the hypothesis of this study is that this combination could focus the immune system on tumor antigens and minimize the aberrant immune activation in normal tissues, consequently reducing the incidence of irAE's (immune related adverse effect). Combination of radiation treatment with Ipilimumab will likely result in better local control, decrease the risk of developing new brain metastases, and improved overall survival. However, the safety profile and toxicities of combining Ipilimumab with brain radiation treatment are unknown. The current phase I study will assess the safety profile of combining different doses of Ipilimumab with standard dose radiation treatment either with WBRT or SRS. The MTD (maximum tolerated dose) will be determined, as well as a recommended phase II trial dose of Ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is >= 18 years
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1.
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
4. Patients must meet the following laboratory criteria:

   * WBC >= 2000/uL
   * ANC >= 1000/uL
   * Platelets >= 75 x 10^3/uL
   * Hemoglobin >= 9 g/dL (>= 80 g/L; may be transfused)
   * AST/ALT <= 2.5 x ULN for patients without liver metastasis
   * AST/ALT <= 5 times for liver metastases
   * Bilirubin <= 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
   * Serum creatinine <= 2.0 x ULN or 24-hour creatinine clearance >= 50 ml/min
   * Total serum calcium (corrected for serum albumin) or ionized calcium >= lower limit of normal (LLN)
   * Serum potassium >= LLN
   * Serum sodium >= LLN
   * Serum albumin >= LLN or 3g/dl
   * Patients with any elevated Alkaline Phosphatase due to bone metastases can be enrolled
5. No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
6. Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
7. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

   * Amenorrhea >= 12 consecutive months without another cause, or
   * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL.
   * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.
   * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.
8. Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized.
9. A pathological diagnosis of melanoma is required, from either the primary or a metastasis. This also includes uveal melanoma.
10. A radiological diagnosis (CT or MRI) of one or more brain metastases is required.
11. Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI CTCAE Version 4.0 grade <= 1.
12. Specific eligibility criteria for the two arms

    * Arm A WBRT and Ipilimumab:

      * Patients have 5 or more brain metastases, or patients have any brain metastases exceeding the limit for SRS (maximum diameter is > 4 cm).
      * OR Patient has only one brain metastasis and completely resected, the resection cavity is > 4 cm in diameter.
    * Arm B SRS and Ipilimumab:

      * Patients have 4 or fewer brain metastases. All the brain metastases are <= 4 cm in diameter.
      * Patients have only one brain metastasis and completely resected, the resection cavity is <= 4 cm in diameter.
      * OR If a patient is found to have progression of brain metastases that exceed 4 cm in diameter based on the MRI scan on the time of SRS procedure, the patient should be re-assigned to WBRT arm or withdrawn from the study. The study PI should be notified.
      * OR If a patient is found to have progression of brain metastases that exceed 4 lesions based on the MRI scan on the time of the SRS procedure, the patient can either be treated with SRS to all the lesions (up to 10 lesions), re-assigned to WBRT arm, or withdrawn from the study per the treating physician. The study PI should be notified.

Exclusion Criteria:

1. Patient with leptomeningeal carcinomatosis.
2. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
3. Major surgery or radiation therapy within 2 weeks of starting the study treatment.
4. If patients are receiving chemotherapy or other investigational drugs, they must be discontinued 4 weeks prior to enrollment.
5. NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
6. Any of the following within the 6 months prior to study drug administration:

   myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism. Patients with known cardiac disease will be required to have an ECHO or MUGA scan at baseline and at the completion of study.
7. Ongoing cardiac dysrhythmias of NCI CTCAE grade >= 2.
8. Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
9. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
10. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
11. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
12. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
13. Concomitant therapy with any of the following: IL-2, interferon, or other non-study immunotherapy regimens, cytotoxic chemotherapy, immunosuppressive agents, vermurafenib, or other investigational therapies.
14. All efforts need to be taken to avoid/minimize the use of cortical steroid during radiation period (1 week prior to start radiation, during radiation, and 1 week after finishing radiation). Any steroid used considered necessary by the treating physician should be closely documented, including medication, route of administration, dose, and duration.
15. Active infection with hepatitis B, or hepatitis C.
16. Patients who had prior brain radiation treatment.
17. Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated basal or squamous cell carcinoma of skin, superficial bladder cancer or carcinoma in situ of cervix, AJCC (version 7.0) stage 0 or I breast cancer, AJCC (version 7.0) stage I, or II prostate cancer.
18. Patients are excluded if they have a history of autoimmune disease, as follows: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Patients with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis) are excluded. Patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy.
19. Patients who are allergic to Ipilimumab.
20. Patients who received ipilimumab before.
21. Patients who are allergic to MRI contrast agent or have contraindication for MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Bafaloukos D, Gogas H. The treatment of brain metastases in melanoma patients. Cancer Treat Rev. 2004 Oct;30(6):515-20. doi: 10.1016/j.ctrv.2004.05.001. PMID 15325032
- [Background] Barth A, Wanek LA, Morton DL. Prognostic factors in 1,521 melanoma patients with distant metastases. J Am Coll Surg. 1995 Sep;181(3):193-201. PMID 7670677
- [Background] Sampson JH, Carter JH Jr, Friedman AH, Seigler HF. Demographics, prognosis, and therapy in 702 patients with brain metastases from malignant melanoma. J Neurosurg. 1998 Jan;88(1):11-20. doi: 10.3171/jns.1998.88.1.0011. PMID 9420067
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] Patchell RA, Tibbs PA, Walsh JW, Dempsey RJ, Maruyama Y, Kryscio RJ, Markesbery WR, Macdonald JS, Young B. A randomized trial of surgery in the treatment of single metastases to the brain. N Engl J Med. 1990 Feb 22;322(8):494-500. doi: 10.1056/NEJM199002223220802. PMID 2405271
- [Background] Andrews DW. Current neurosurgical management of brain metastases. Semin Oncol. 2008 Apr;35(2):100-7. doi: 10.1053/j.seminoncol.2007.12.003. PMID 18396195
- [Background] Thomas SS, Dunbar EM. Modern multidisciplinary management of brain metastases. Curr Oncol Rep. 2010 Jan;12(1):34-40. doi: 10.1007/s11912-009-0073-8. PMID 20425606
- [Background] CHU FC, HILARIS BB. Value of radiation theray in the management of intracranial metastases. Cancer. 1961 May-Jun;14:577-81. doi: 10.1002/1097-0142(199005/06)14:33.0.co;2-f. No abstract available. PMID 13693470
- [Background] Expert Panel on Radiation Oncology-Brain Metastases; Videtic GM, Gaspar LE, Aref AM, Germano IM, Goldsmith BJ, Imperato JP, Marcus KJ, McDermott MW, McDonald MW, Patchell RA, Robins HI, Rogers CL, Suh JH, Wolfson AH, Wippold FJ 2nd. American College of Radiology appropriateness criteria on multiple brain metastases. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):961-5. doi: 10.1016/j.ijrobp.2009.07.1720. No abstract available. PMID 19857783
- [Background] DiLuna ML, King JT Jr, Knisely JP, Chiang VL. Prognostic factors for survival after stereotactic radiosurgery vary with the number of cerebral metastases. Cancer. 2007 Jan 1;109(1):135-45. doi: 10.1002/cncr.22367. PMID 17133440
- [Background] Manon R, O'Neill A, Knisely J, Werner-Wasik M, Lazarus HM, Wagner H, Gilbert M, Mehta M; Eastern Cooperative Oncology Group. Phase II trial of radiosurgery for one to three newly diagnosed brain metastases from renal cell carcinoma, melanoma, and sarcoma: an Eastern Cooperative Oncology Group study (E 6397). J Clin Oncol. 2005 Dec 1;23(34):8870-6. doi: 10.1200/JCO.2005.01.8747. PMID 16314647
- [Background] Mathieu D, Kondziolka D, Cooper PB, Flickinger JC, Niranjan A, Agarwala S, Kirkwood J, Lunsford LD. Gamma knife radiosurgery for malignant melanoma brain metastases. Clin Neurosurg. 2007;54:241-7. No abstract available. PMID 18504926
- [Background] Clarke JW, Register S, McGregor JM, Grecula JC, Mayr NA, Wang JZ, Li K, Gupta N, Kendra KL, Olencki TE, Cavaliere R, Sarkar A, Lo SS. Stereotactic radiosurgery with or without whole brain radiotherapy for patients with a single radioresistant brain metastasis. Am J Clin Oncol. 2010 Feb;33(1):70-4. doi: 10.1097/COC.0b013e31819ccc8c. PMID 19652578
- [Background] Order SE, Hellman S, Von Essen CF, Kligerman MM. Improvement in quality of survival following whole-brain irradiation for brain metastasis. Radiology. 1968 Jul;91(1):149-53. doi: 10.1148/91.1.149. No abstract available. PMID 4172540
- [Background] Khuntia D, Brown P, Li J, Mehta MP. Whole-brain radiotherapy in the management of brain metastasis. J Clin Oncol. 2006 Mar 10;24(8):1295-304. doi: 10.1200/JCO.2005.04.6185. PMID 16525185
- [Background] Patchell RA, Regine WF. The rationale for adjuvant whole brain radiation therapy with radiosurgery in the treatment of single brain metastases. Technol Cancer Res Treat. 2003 Apr;2(2):111-5. doi: 10.1177/153303460300200206. PMID 12680791
- [Background] Borgelt B, Gelber R, Larson M, Hendrickson F, Griffin T, Roth R. Ultra-rapid high dose irradiation schedules for the palliation of brain metastases: final results of the first two studies by the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 1981 Dec;7(12):1633-8. doi: 10.1016/0360-3016(81)90184-x. No abstract available. PMID 6174490
- [Background] Chatani M, Matayoshi Y, Masaki N, Inoue T. Radiation therapy for brain metastases from lung carcinoma. Prospective randomized trial according to the level of lactate dehydrogenase. Strahlenther Onkol. 1994 Mar;170(3):155-61. PMID 8160096
- [Background] Haie-Meder C, Pellae-Cosset B, Laplanche A, Lagrange JL, Tuchais C, Nogues C, Arriagada R. Results of a randomized clinical trial comparing two radiation schedules in the palliative treatment of brain metastases. Radiother Oncol. 1993 Feb;26(2):111-6. doi: 10.1016/0167-8140(93)90091-l. PMID 7681997
- [Background] Harwood AR, Simson WJ. Radiation therapy of cerebral metastases: a randomized prospective clinical trial. Int J Radiat Oncol Biol Phys. 1977 Nov-Dec;2(11-12):1091-4. doi: 10.1016/0360-3016(77)90114-6. No abstract available. PMID 74375
- [Background] Kurtz JM, Gelber R, Brady LW, Carella RJ, Cooper JS. The palliation of brain metastases in a favorable patient population: a randomized clinical trial by the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 1981 Jul;7(7):891-5. doi: 10.1016/0360-3016(81)90005-5. No abstract available. PMID 6171553
- [Background] Murray KJ, Scott C, Greenberg HM, Emami B, Seider M, Vora NL, Olson C, Whitton A, Movsas B, Curran W. A randomized phase III study of accelerated hyperfractionation versus standard in patients with unresected brain metastases: a report of the Radiation Therapy Oncology Group (RTOG) 9104. Int J Radiat Oncol Biol Phys. 1997 Oct 1;39(3):571-4. doi: 10.1016/s0360-3016(97)00341-6. PMID 9336134
- [Background] Davey P, Hoegler D, Ennis M, Smith J. A phase III study of accelerated versus conventional hypofractionated whole brain irradiation in patients of good performance status with brain metastases not suitable for surgical excision. Radiother Oncol. 2008 Aug;88(2):173-6. doi: 10.1016/j.radonc.2008.05.020. Epub 2008 Jun 12. PMID 18555546
- [Background] Mehta MP, Tsao MN, Whelan TJ, Morris DE, Hayman JA, Flickinger JC, Mills M, Rogers CL, Souhami L. The American Society for Therapeutic Radiology and Oncology (ASTRO) evidence-based review of the role of radiosurgery for brain metastases. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):37-46. doi: 10.1016/j.ijrobp.2005.05.023. PMID 16111570
- [Background] Meyners T, Heisterkamp C, Kueter JD, Veninga T, Stalpers LJ, Schild SE, Rades D. Prognostic factors for outcomes after whole-brain irradiation of brain metastases from relatively radioresistant tumors: a retrospective analysis. BMC Cancer. 2010 Oct 26;10:582. doi: 10.1186/1471-2407-10-582. PMID 20977700
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Pirzkall A, Debus J, Lohr F, Fuss M, Rhein B, Engenhart-Cabillic R, Wannenmacher M. Radiosurgery alone or in combination with whole-brain radiotherapy for brain metastases. J Clin Oncol. 1998 Nov;16(11):3563-9. doi: 10.1200/JCO.1998.16.11.3563. PMID 9817276
- [Background] Sheehan JP, Sun MH, Kondziolka D, Flickinger J, Lunsford LD. Radiosurgery in patients with renal cell carcinoma metastasis to the brain: long-term outcomes and prognostic factors influencing survival and local tumor control. J Neurosurg. 2003 Feb;98(2):342-9. doi: 10.3171/jns.2003.98.2.0342. PMID 12593621
- [Background] Powell JW, Chung CT, Shah HR, Canute GW, Hodge CJ, Bassano DA, Liu L, Mitchell L, Hahn SS. Gamma Knife surgery in the management of radioresistant brain metastases in high-risk patients with melanoma, renal cell carcinoma, and sarcoma. J Neurosurg. 2008 Dec;109 Suppl:122-8. doi: 10.3171/JNS/2008/109/12/S19. PMID 19123898
- [Background] Lo SS, Clarke JW, Grecula JC, McGregor JM, Mayr NA, Cavaliere R, Kendra KL, Gupta N, Wang JZ, Sarkar A, Olencki TE. Stereotactic radiosurgery alone for patients with 1-4 radioresistant brain metastases. Med Oncol. 2011 Dec;28 Suppl 1:S439-44. doi: 10.1007/s12032-010-9670-5. Epub 2010 Sep 3. PMID 20814764
- [Background] Nagorsen D, Scheibenbogen C, Marincola FM, Letsch A, Keilholz U. Natural T cell immunity against cancer. Clin Cancer Res. 2003 Oct 1;9(12):4296-303. PMID 14555498
- [Background] Clemente CG, Mihm MC Jr, Bufalino R, Zurrida S, Collini P, Cascinelli N. Prognostic value of tumor infiltrating lymphocytes in the vertical growth phase of primary cutaneous melanoma. Cancer. 1996 Apr 1;77(7):1303-10. doi: 10.1002/(SICI)1097-0142(19960401)77:73.0.CO;2-5. PMID 8608507
- [Background] Hakansson A, Gustafsson B, Krysander L, Hakansson L. Tumour-infiltrating lymphocytes in metastatic malignant melanoma and response to interferon alpha treatment. Br J Cancer. 1996 Sep;74(5):670-6. doi: 10.1038/bjc.1996.420. PMID 8845294
- [Background] Mihm MC Jr, Clemente CG, Cascinelli N. Tumor infiltrating lymphocytes in lymph node melanoma metastases: a histopathologic prognostic indicator and an expression of local immune response. Lab Invest. 1996 Jan;74(1):43-7. PMID 8569196
- [Background] Moschos SJ, Edington HD, Land SR, Rao UN, Jukic D, Shipe-Spotloe J, Kirkwood JM. Neoadjuvant treatment of regional stage IIIB melanoma with high-dose interferon alfa-2b induces objective tumor regression in association with modulation of tumor infiltrating host cellular immune responses. J Clin Oncol. 2006 Jul 1;24(19):3164-71. doi: 10.1200/JCO.2005.05.2498. PMID 16809739
- [Background] Peggs KS, Quezada SA, Korman AJ, Allison JP. Principles and use of anti-CTLA4 antibody in human cancer immunotherapy. Curr Opin Immunol. 2006 Apr;18(2):206-13. doi: 10.1016/j.coi.2006.01.011. Epub 2006 Feb 7. PMID 16464564
- [Background] Tarhini AA, Iqbal F. CTLA-4 blockade: therapeutic potential in cancer treatments. Onco Targets Ther. 2010 Jun 24;3:15-25. doi: 10.2147/ott.s4833. PMID 20616954
- [Background] Robert C, Ghiringhelli F. What is the role of cytotoxic T lymphocyte-associated antigen 4 blockade in patients with metastatic melanoma? Oncologist. 2009 Aug;14(8):848-61. doi: 10.1634/theoncologist.2009-0028. Epub 2009 Aug 1. PMID 19648604
- [Background] Read S, Malmstrom V, Powrie F. Cytotoxic T lymphocyte-associated antigen 4 plays an essential role in the function of CD25(+)CD4(+) regulatory cells that control intestinal inflammation. J Exp Med. 2000 Jul 17;192(2):295-302. doi: 10.1084/jem.192.2.295. PMID 10899916
- [Background] Kaehler KC, Piel S, Livingstone E, Schilling B, Hauschild A, Schadendorf D. Update on immunologic therapy with anti-CTLA-4 antibodies in melanoma: identification of clinical and biological response patterns, immune-related adverse events, and their management. Semin Oncol. 2010 Oct;37(5):485-98. doi: 10.1053/j.seminoncol.2010.09.003. PMID 21074064
- [Background] Morse MA. Technology evaluation: ipilimumab, Medarex/Bristol-Myers Squibb. Curr Opin Mol Ther. 2005 Dec;7(6):588-97. PMID 16370382
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Weber JS, O'Day S, Urba W, Powderly J, Nichol G, Yellin M, Snively J, Hersh E. Phase I/II study of ipilimumab for patients with metastatic melanoma. J Clin Oncol. 2008 Dec 20;26(36):5950-6. doi: 10.1200/JCO.2008.16.1927. Epub 2008 Nov 17. PMID 19018089
- [Background] Schartz NE, Farges C, Madelaine I, Bruzzoni H, Calvo F, Hoos A, Lebbe C. Complete regression of a previously untreated melanoma brain metastasis with ipilimumab. Melanoma Res. 2010 Jun;20(3):247-50. doi: 10.1097/CMR.0b013e3283364a37. PMID 20216240
- [Background] Hodi FS, Oble DA, Drappatz J, Velazquez EF, Ramaiya N, Ramakrishna N, Day AL, Kruse A, Mac Rae S, Hoos A, Mihm M. CTLA-4 blockade with ipilimumab induces significant clinical benefit in a female with melanoma metastases to the CNS. Nat Clin Pract Oncol. 2008 Sep;5(9):557-61. doi: 10.1038/ncponc1183. Epub 2008 Jul 29. PMID 18665147
- [Background] Pilones KA, Kawashima N, Yang AM, Babb JS, Formenti SC, Demaria S. Invariant natural killer T cells regulate breast cancer response to radiation and CTLA-4 blockade. Clin Cancer Res. 2009 Jan 15;15(2):597-606. doi: 10.1158/1078-0432.CCR-08-1277. PMID 19147765
- [Background] Jaber SH, Cowen EW, Haworth LR, Booher SL, Berman DM, Rosenberg SA, Hwang ST. Skin reactions in a subset of patients with stage IV melanoma treated with anti-cytotoxic T-lymphocyte antigen 4 monoclonal antibody as a single agent. Arch Dermatol. 2006 Feb;142(2):166-72. doi: 10.1001/archderm.142.2.166. PMID 16490844
- [Background] Robinson MR, Chan CC, Yang JC, Rubin BI, Gracia GJ, Sen HN, Csaky KG, Rosenberg SA. Cytotoxic T lymphocyte-associated antigen 4 blockade in patients with metastatic melanoma: a new cause of uveitis. J Immunother. 2004 Nov-Dec;27(6):478-9. doi: 10.1097/00002371-200411000-00008. PMID 15534492
- [Background] Hodi FS, Butler M, Oble DA, Seiden MV, Haluska FG, Kruse A, Macrae S, Nelson M, Canning C, Lowy I, Korman A, Lautz D, Russell S, Jaklitsch MT, Ramaiya N, Chen TC, Neuberg D, Allison JP, Mihm MC, Dranoff G. Immunologic and clinical effects of antibody blockade of cytotoxic T lymphocyte-associated antigen 4 in previously vaccinated cancer patients. Proc Natl Acad Sci U S A. 2008 Feb 26;105(8):3005-10. doi: 10.1073/pnas.0712237105. Epub 2008 Feb 19. PMID 18287062
- [Background] Downey SG, Klapper JA, Smith FO, Yang JC, Sherry RM, Royal RE, Kammula US, Hughes MS, Allen TE, Levy CL, Yellin M, Nichol G, White DE, Steinberg SM, Rosenberg SA. Prognostic factors related to clinical response in patients with metastatic melanoma treated by CTL-associated antigen-4 blockade. Clin Cancer Res. 2007 Nov 15;13(22 Pt 1):6681-8. doi: 10.1158/1078-0432.CCR-07-0187. Epub 2007 Nov 2. PMID 17982122
- [Background] Korn EL, Liu PY, Lee SJ, Chapman JA, Niedzwiecki D, Suman VJ, Moon J, Sondak VK, Atkins MB, Eisenhauer EA, Parulekar W, Markovic SN, Saxman S, Kirkwood JM. Meta-analysis of phase II cooperative group trials in metastatic stage IV melanoma to determine progression-free and overall survival benchmarks for future phase II trials. J Clin Oncol. 2008 Feb 1;26(4):527-34. doi: 10.1200/JCO.2007.12.7837. PMID 18235113
- [Background] Chapman PB, Einhorn LH, Meyers ML, Saxman S, Destro AN, Panageas KS, Begg CB, Agarwala SS, Schuchter LM, Ernstoff MS, Houghton AN, Kirkwood JM. Phase III multicenter randomized trial of the Dartmouth regimen versus dacarbazine in patients with metastatic melanoma. J Clin Oncol. 1999 Sep;17(9):2745-51. doi: 10.1200/JCO.1999.17.9.2745. PMID 10561349
- [Background] Middleton MR, Lorigan P, Owen J, Ashcroft L, Lee SM, Harper P, Thatcher N. A randomized phase III study comparing dacarbazine, BCNU, cisplatin and tamoxifen with dacarbazine and interferon in advanced melanoma. Br J Cancer. 2000 Mar;82(6):1158-62. doi: 10.1054/bjoc.1999.1056. PMID 10735499
- [Background] Bedikian AY, Millward M, Pehamberger H, Conry R, Gore M, Trefzer U, Pavlick AC, DeConti R, Hersh EM, Hersey P, Kirkwood JM, Haluska FG; Oblimersen Melanoma Study Group. Bcl-2 antisense (oblimersen sodium) plus dacarbazine in patients with advanced melanoma: the Oblimersen Melanoma Study Group. J Clin Oncol. 2006 Oct 10;24(29):4738-45. doi: 10.1200/JCO.2006.06.0483. Epub 2006 Sep 11. PMID 16966688
- [Background] van Elsas A, Hurwitz AA, Allison JP. Combination immunotherapy of B16 melanoma using anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) and granulocyte/macrophage colony-stimulating factor (GM-CSF)-producing vaccines induces rejection of subcutaneous and metastatic tumors accompanied by autoimmune depigmentation. J Exp Med. 1999 Aug 2;190(3):355-66. doi: 10.1084/jem.190.3.355. PMID 10430624
- [Background] Suh JH, Videtic GM, Aref AM, Germano I, Goldsmith BJ, Imperato JP, Marcus KJ, McDermott MW, McDonald MW, Patchell RA, Robins HI, Rogers CL, Wolfson AH, Wippold FJ 2nd, Gaspar LE. ACR Appropriateness Criteria: single brain metastasis. Curr Probl Cancer. 2010 May-Jun;34(3):162-74. doi: 10.1016/j.currproblcancer.2010.04.003. PMID 20541055
- [Background] Shaw E, Scott C, Souhami L, Dinapoli R, Kline R, Loeffler J, Farnan N. Single dose radiosurgical treatment of recurrent previously irradiated primary brain tumors and brain metastases: final report of RTOG protocol 90-05. Int J Radiat Oncol Biol Phys. 2000 May 1;47(2):291-8. doi: 10.1016/s0360-3016(99)00507-6. PMID 10802351
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Derived] Williams NL, Wuthrick EJ, Kim H, Palmer JD, Garg S, Eldredge-Hindy H, Daskalakis C, Feeney KJ, Mastrangelo MJ, Kim LJ, Sato T, Kendra KL, Olencki T, Liebner DA, Farrell CJ, Evans JJ, Judy KD, Andrews DW, Dicker AP, Werner-Wasik M, Shi W. Phase 1 Study of Ipilimumab Combined With Whole Brain Radiation Therapy or Radiosurgery for Melanoma Patients With Brain Metastases. Int J Radiat Oncol Biol Phys. 2017 Sep 1;99(1):22-30. doi: 10.1016/j.ijrobp.2017.05.028. Epub 2017 May 26. PMID 28816150
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Started | 6 | 11
Completed | 5 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery) | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 8 | 9
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 11 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Ipilimumab
Description: (MTD) when combined with WBRT or SRS, defined as the last dose studied or the previous dose, based on clinical judgment of the degree of toxicity seen at the last dose
Time Frame: 30 days following the completion of radiation therapy
Measure: Number; unit: mg/kg
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 5 | 11
mg/kg | 3 | 10

2. Secondary Outcome: Rate of Developing New Brain Metastases in Each Arm
Time Frame: Up to 5 years
Population: Of the enrolled participants, only 7 developed new Brain Metastases (BMs) and were included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 1 | 6
months | 8.2 [8.2 to 8.2] | 1.9 [0.97 to 8.2]

3. Secondary Outcome: Number of Subjects With Response of Extracranial Disease
Description: Extracranial disease is assessed through repeated computed tomography of the chest, abdomen, and pelvis. The purpose of this scan is to determine if there is any evidence of disease outside of the brain.
Time Frame: Up to 5 years
Population: Of the enrolled participants, only 4 out of 5 participants on Arm A and 9 out of 11 participants on Arm B had Extracranial Disease. Only these participants were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 4 | 9
Participants | 0 | 5

4. Secondary Outcome: Overall Survival (OS) Rate
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 5 | 11
months | 8 [3.5 to 24.1] | 10.5 [1.8 to 36.8]

5. Secondary Outcome: Number of Patients With Progression Free Survival (PFS) Rate
Description: PFS rate based on Response Evaluation Criteria in Solid Tumors (RECIST) and immune-related response criteria (irRC) criteria based on the brain MRI and systematic assessment by the treating physician
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 5 | 11
Participants | 3 | 3

6. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Time Frame: 4 weeks following the last dose of ipilimumab
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
Number analyzed (Participants) | 5 | 11
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: 30 days after completion of radiation therapy (RT)
Arm/Group | Arm A (Ipilimumab and Whole Brain Radiation Therapy) | Arm B (Ipilimumab and Stereotactic Radiosurgery)
All-Cause Mortality (participants affected / at risk) | 3/5 | 3/11
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/11
Other Adverse Events (participants affected / at risk) | 2/5 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ipilimumab and Whole Brain Radiation Therapy) (N=5) | Arm B (Ipilimumab and Stereotactic Radiosurgery) (N=11)
diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ipilimumab and Whole Brain Radiation Therapy) (N=5) | Arm B (Ipilimumab and Stereotactic Radiosurgery) (N=11)
headache (General disorders) | 2 | 4
fatigue (General disorders) | 1 | 1
Changes in Hearing (Ear and labyrinth disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3
Anoerexia (Metabolism and nutrition disorders) | 2 | 1
hot flashes (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Vision Changes (Eye disorders) | 0 | 1
hypertension (Vascular disorders) | 2 | 0
Alopecia (General disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Dizziness (General disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Depression (General disorders) | 0 | 1
Lipase Increase (Hepatobiliary disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Facial Palsy (Nervous system disorders) | 0 | 1
Pleural effusion (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes